CLINICAL TRIAL: NCT01206712
Title: Beta Cell Relieving and Cardiovascular Protective Effects of LANTUS Treatment in Type 2 Diabetes Patients - Investigation on Postprandial Excursions of Proinsulin and PAI-1 Levels
Brief Title: Beta Cell Relieving and Cardiovascular Protective Effects of LANTUS Treatment in Type 2 Diabetes Patients
Status: Completed | Type: Observational
Sponsor: ikfe-CRO GmbH (Industry)
Collaborators: Sanofi (Industry); IKFE Institute for Clinical Research and Development (Other)
Responsible Party: Prof. Dr. Thomas Forst, IKFE Institute for Clinical Research and Development
Other Study IDs: SAN-FORST-001
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2010-09-22 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus Type 2; insulin glargine; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- T2DM patients treated with LANTUS + MET: T2DM patients treated with LANTUS + Metformin(MET) in their routine antidiabetic therapy. These patients do not receive any study specific medication.
- T2DM patients treated with SU + MET: T2DM patients treated with Sulfonylurea (SU) + Metformin(MET)in their routine antidiabetic therapy. These patients do not receive any study specific medication.
- T2DM patients treated with DPP-4 + MET: T2DM patients treated with Dipeptidylpeptidase 4 inhibitors (DPP-4) + Metformin(MET) in their routine antidiabetic therapy. These patients do not receive any study specific medication.
- Healthy subjects: healthy volunteres who do not receive any antidiabetic medication in their routine therapie.

SUMMARY:
The purpose of this phase IV clinical trial is to investigate the effect of Insulin glargine + metformin treatment vs. sulfonylurea + metformin treatment vs. DPP-4 + metformin treatment vs. healthy volunteers on ß-cell function after the uptake of a standardized meal.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus is a progressive disease characterised by a steady loss of beta cell function and an increase in the proinsulin/insulin ratio. During the recent years intact proinsulin has been the topic of interest in numerous preclinical and clinical studies in patients with type 2 diabetes mellitus. Intact proinsulin was confirmed as a marker of functional beta cell failure and as a predictor of increased beta cell loss due to apoptosis and/or diminished neogenesis.

A number of population based studies showed that intact proinsulin is a strong predictor of coronary heart disease in diabetic, and in non-diabetic patients. In a clinical trial investigating human proinsulin as a therapeutic approach for the treatment of diabetes mellitus an eight fold increase in CVD was found during treatment with human proinsulin compared to human regular insulin, indicating a thrombo-embolic potential of intact proinsulin. In a recent investigation an association could be confirmed between increased proinsulin plasma concentrations and the severity of angiographical characterised CHD.

Even the exact mechanism how proinsulin is involved in the pathogenesis of atherosclerosis is not completely recognized, it was already shown that PAI-1 activity increases after proinsulin administration in vitro, and there is increasing evidence that the atherogenic effects of proinsulin might be linked to increasing plasminogen activator inhibitor-1 (PAI-1) levels with subsequent inhibition of fibrinolysis and an augmented thrombogenic potency.

Treatment with sulfonylurea increases intact proinsulin secretion, and in a couple of studies, sulfonylurea treatment was found to be associated with an increased cardiovascular risk. In contrast, several studies have shown that after the introduction of insulin treatment in type 2 diabetic patients intact proinsulin levels and plasma PAI 1 levels decline, indicating not only beta cell protection, but also antiatherogenic properties of insulin. In a recent study, we have shown that treatment with basal insulin in combination with metformin effectively reduces intact proinsulin levels, and that insulin glargine is superior to NPH insulin in controlling postprandial release of intact proinsulin over an entire day.

Recently a new therapeutic concept using DPP IV inhibitors in combination with metformin has been introduced in the treatment of type 2 diabetic patients. There is some evidence that, in the beta cell, DPP IV Inhibitors might improve the conversion of intact Proinsulin into Insulin and C-peptide and thereby reduce circulating intact proinsulin levels. Since the number of type 2 diabetic patients treated with DPP-IV inhibitors is steadily increasing, there is a need to generate more data on the postprandial release of intact proinsulin in patients treated with DPP-IV inhibitors compared to Insulin or sulfonylurea treatment.

The rationale of the study is to investigate the effect of glargine and metformin treatment compared to sulfonylurea and metformin treatment and compared to DPP-4 inhibitor and metformin treatment on postprandial intact proinsulin release and postprandial PAI-1 levels. Accompanying a comparison of postprandial intact proinsulin release and the time course of postprandial PAI-levels in between all three antidiabetic treatment groups and a non-diabetic control group will be performed as well.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria - applicable for T2DM group only:

   1.1. Type 2 diabetes mellitus 1.2. Duration of T2DM between 3 and 15 years inclusively 1.3. HbA1c up to 7.5% inclusively 1.4. Treated with LANTUS+MET (Group LANTUS+MET) or SU+MET (Group SU+MET) or DPP-4+MET (Group DPP-4+MET) respectively during the past 6 months before entering the study 1.5. Treated on a stable antidiabetic dosage during the past 3 months before entering the study
2. Inclusion criteria - applicable for healthy subject only:

   2.1. Fasting blood glucose £ 100 mg/dl (5.6 mmol/l) 2.2. Oral Glucose Tolerance Test (OGTT) revealed no IGT or DM

   Inclusion criteria - applicable for all subjects:
3. Age of 40-75 years inclusively
4. BMI between 20 and 35 kg/m2 inclusively
5. Patient informed consent

Exclusion Criteria:

1. Exclusion criteria - applicable for T2DM group only:

   1.1. Type 1 diabetes mellitus 1.2. Treatment with any other insulin than LANTUS during the past 6 months in Group LANTUS+MET or with any kind of insulin during the past 3 months in Group SU+MET or Group DPP-4+MET before entering the study 1.3. Treatment with any kind of OAD except MET during the past 6 months in Group LANTUS+MET or with any kind of OAD except MET+SU during the past 3 months in Group SU+MET or with any kind of OAD except DPP-4+SU during the past 3 months in Group DPP-4+MET before entering the study 1.4. Major micro- or macro vascular complications as judged by the investigator
2. Exclusion criteria - applicable for healthy subject only:

   2.1. Type 1 or type 2 diabetes mellitus (checked by oGTT) 2.2. Impaired Glucose Tolerance (IGT, checked by oGTT) 2.3. Impaired Fasting Glucose (IFG, checked by oGTT)

   Exclusion criteria - applicable for all subjects:
3. History of drug or alcohol abuse within the last five years prior to screening
4. History of severe or multiple allergies
5. Treatment with any other investigational drug within 3 months prior to screening
6. Progressive fatal disease
7. Known psychiatric illness
8. History of significant cardiovascular, respiratory, gastrointestinal, hepatic (ALAT and/or ASAT > 3 times the normal reference range), renal (creatinine > 1.1 mg/dl in women and > 1.5 mg/dl in men), neurological, psychiatric and/or haematological disease as judged by the investigator
9. Pregnancy or breast feeding
10. Sexually active women of childbearing potential not consistently and correctly practicing birth control by implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence or vasectomised partner
11. Lack of compliance or other similar reason, that according to investigator, precludes satisfactory participation in the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Group 1 (n=20): Healthy subjects
  * Group 2 (n=20): T2DM patients treated with continuous SU + MET therapy as individually prescriped by the primary care physicians
  * Group 3 (n=20): T2DM patients treated with continuous LANTUS + MET therapy as individually prescriped by the primary care physicians
  * Group 4 (n=20): T2DM patients treated with continuous DPP-4 + MET therapy as individually prescriped by the primary care physicians
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-11; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Investigation of ß-cell function via comparison of AUC0-300 minutes of intact Proinsulin in T2DM patients treated with LANTUS + Metformin (MET) vs. T2DM patients treated with Sulfonylurea (SU) + Metformin | 0-300 minutes after standardized meal
  Comparison of AUC0-300 min [intact Proinsulin] between T2DM patients treated with LANTUS + Metformin and T2DM patients treated with Sulfonylurea + MET after uptake of standardized meal

SECONDARY OUTCOMES:
Investigation of insulin, intact proinsulin, glucose and PAI-1 levels over a 5 h period after uptake of a standardized meal comparing four different population groups | 0-300 minutes after standardized meal
  Comparison of the AUC0-300 of intact proinsulin between each of the 4 treatment groups with the exception of T2DM patients treated with LANTUS + MET and T2DM patients treated with SU + MET after uptake of a standardized meal.
  Comparison of the AUC0-300 for insulin, the AUC0-300 and the AUC0-180 for blood glucose, the mean maximum levels of intact proinsulin, insulin and BG, and the PAI-1 level excursion at the time points 0, 150 and 300 min between each of the 4 treatment groups.
  Comparison of the change in the insulin/intact proinsulin ratio between each of the 4 treatment groups

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, Prof. MD, Principal Investigator — IKFE Institute for Clinical Research and Development
Locations (1):
- IKFE Institute for Clinical Research and Development, Mainz, Germany